CLINICAL TRIAL: NCT04219163
Title: Chimeric Antigen Receptor T-cells for The Treatment of Acute Myeloid Leukemia Expressing CLL-1 Antigen
Brief Title: Chimeric Antigen Receptor T-cells for The Treatment of AML Expressing CLL-1 Antigen
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: The Methodist Hospital Research Institute (Other); Center for Cell and Gene Therapy, Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, LaQuisa Hill, Assistant Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-43516-CARMEN; 52988-C1 (Other Grant/Funding Number: CPRIT)
Record Dates: First submitted 2020-01-03; First posted 2020-01-06 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-08

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- CLL-1.CAR (Experimental): Group A
  Interventions: Biological: CLL-1.CAR T cells

INTERVENTIONS:
Biological: CLL-1.CAR T cells — Dose escalation study with 3 dose levels:
  DL1: 1x10^7 cells/m2, DL2: 3x10^7 cells/m2, DL3: 1x10^8 cells/m2
  If excessive dose limiting toxicity attributed to the product occurs at dose level one, we will request permission from FDA to treat at dose level -1: 5×10^6 cells/m2

SUMMARY:
Patients eligible for this study have a type of blood cancer Acute Myeloid Leukemia (AML) which has come back or has not gone away after treatment.

The body has different ways of fighting disease and infection, and this research study combines two different ways of fighting cancer with antibodies and T cells with the hope that they will work together. T cells (also called T lymphocytes) are special infection-fighting blood cells that can kill other cells including tumor cells. Antibodies are types of proteins that protect the body from bacterial and other infectious diseases. Both antibodies and T cells have been used to treat patients with cancers; they have shown promise, but have not been strong enough to cure most patients when used alone.

T lymphocytes can kill tumor cells but there normally are not enough of them to kill all the tumor cells. Some researchers have taken T cells from a person's blood, grown more of them in the laboratory and then given them back to the person. The antibody used in this study targets CLL-1. This antibody sticks to AML cells because of a substance (protein) on the outside of these cells called CLL-1. For this study, the antibody to CLL-1 has been changed so that instead of floating free in the blood, it is now joined to the T cells. When T-cells contain an antibody that is joined to them, they are called chimeric antigen receptor T-cells or CAR-T cells.

In the laboratory, the investigators have also found that T cells work better if proteins that stimulate T cells are also added, such as one called CD28. Adding the CD28 makes the cells grow better and last longer in the body, thus giving the cells a better chance of killing the leukemia or lymphoma cells. In this study we are going to attach the CLL-1 chimeric receptor that has CD28 added to it to the patient's T cells. We will then test how long the cells last.

These CLL-1 chimeric antigen receptor T cells with CD28 are investigational products not approved by the Food and Drug Administration.

DETAILED DESCRIPTION:
To make the CLL1-CD28 chimeric antigen receptor T cells, the investigators will collect the patient's blood and stimulate them with growth factors to make the cells grow. To get the CLL-1 antibody and CD28 to attach to the surface of the T cell, we put the antibody gene into the T cell. This is done using a virus called a retrovirus that has been made for this study and will carry the antibody gene into the T cell. This virus also helps investigators find the T cells in the patient's blood after they are injected. Because the patient will receive cells with a new gene in them the patient will be followed for a total of 15 years to see if there are any long term side effects of gene transfer.

When the patient enrolls on this study, the patient will be assigned a dose of CLL-1 chimeric antigen receptor- T cells. Several studies suggest that the T cells that we give to the patient need room to be able to grow and work well and that this may not happen if there are too many other T cells already circulating in the patient's body. Because of that, the patient will receive two chemotherapy medications before receiving the CLL-1 chimeric antigen receptor- T cells.

One medication is called cyclophosphamide and and the other will be either fludarabine or clofarabine. The patient will receive 3 daily doses of each drug, finishing at least one day before receiving the chimeric antigen receptor- T cells. These drugs will lower the numbers of the patient's T cells before we give them the CLL-1 chimeric antigen receptor T cells and will also help lower the number of other cells that may block the chimeric antigen receptor-T cells from working well. Although we do not expect any effect on the patient's cancer with the doses that will be received, these drugs are part of many treatment plans that are used to treat leukemia.

Patients will be given an injection of cells into the vein through an IV at the assigned dose at a minimum of 24 hours after completing the chemotherapy medications. The injection will take from 1 to 10 minutes. Before patients receive the injection, they may be given a dose of Benadryl and Tylenol. The treatment will be given by the Center for Cell and Gene Therapy at Texas Children's Hospital or Houston Methodist Hospital.

If the patient is one of the first set of enrolled patients, they will be admitted as an inpatient for at least 72 hours so that the doctor and nurses can watch them closely in case any potential side effects occur following infusion. After discharge from the hospital you will be followed closely in the clinic, and will have to remain in the Houston area for at least 4 weeks after the infusion. If patients have any side effects, they may have to be admitted to the hospital for evaluation and management. If after a 4 week evaluation period following the infusion, the patient has achieved a complete response, his/her cancer doctors may decide if you should go on to have a bone marrow transplant, at which time the patient will be removed from the treatment portion of the study

BEFORE BEING TREATED, PATIENTS WILL RECEIVE A SERIES OF STANDARD MEDICAL TESTS:

* Physical exam and History
* Blood tests to measure blood cells, kidney and liver function
* Pregnancy test for female patients who are of child bearing potential -Measurements of your tumor by bone marrow studies
* Imaging such as PET scans, CT scans or MRIs will be obtained if needed

PATIENTS WILL RECEIVE STANDARD MEDICAL TESTS DURING TREATMENT AND AFTER:

* Physical exams and History
* Blood tests to measure blood cells, kidney and liver function
* Measurements of your tumor by bone marrow studies 4-6 weeks after the infusion, possibly 12 weeks after the infusion and then per standard of care.
* Imaging such as PET scans, CT scans or MRIs will be obtained if needed 4-6 weeks following the infusion

To learn more about the way the CLL-1 chimeric receptor-T cells are working and how long they last in the body, extra blood will be drawn. The total amount on any day is about 10 teaspoons (50 mL) or no more than 3 mL per 2.2 pounds body weight in children. This amount is considered safe but may be lowered if you are anemic. This blood may be taken from a central line if you have one. Blood will be taken before the chemotherapy drugs, before the T cell infusion, several hours after the T cell infusion, at 1 week, 2 weeks, 3 weeks, 4 weeks, 6 weeks, and 8 weeks after the infusion, at 3 months, 6 months, 9 months, at 1 year, every 6 months for 4 years, then yearly for a total of 15 years.

If patients have a bone marrow exam while they are on this study, we may ask to have a sample of bone marrow to look for CLL-1 chimeric receptor- T cells.

If a patient decides to withdraw at any time during the study, both samples and data collected during his/her participation will be kept.

ELIGIBILITY:
PROCUREMENT

Inclusion Criteria:

1. Diagnosis of primary refractory or relapsed Acute Myeloid Leukemia (AML) with the exception of acute promyelocytic leukemia (APL) AND suitable for consideration of allogeneic Hematopoietic Stem Cell Transplant with confirmation of an identified eligible donor by a FACT accredited transplant center
2. CLL-1 positive tumor with at least 30% CLL-1 blasts by flow cytometry or immunohistochemistry (tissue) assessed by a CLIA certified Flow Cytometry/Pathology laboratory
3. Age ≤75 years NOTE: The first six (6) patients treated on the study will be adults (≥18 yrs of age).
4. Hgb ≥ 7.0 g/dL(can be transfused)
5. Life expectancy greater than 12 wks
6. If apheresis required to collect blood

   * PT and APTT <1.5x ULN
   * Serum Creatinine < 1.5 x ULN
   * AST < 1.5 x ULN
7. Informed consent

Exclusion Criteria:

1. Diagnosis of acute promyelocytic leukemia (APL)
2. Active infection (bacterial, fungal or viral) requiring ongoing treatment without improvement.
3. Active infection with HIV or HTLV (results may be pending)
4. Active second cancer (except non-melanoma skin cancer or in situ breast cancer or cervix cancer)or other cancer treated ≤ 2 years prior to enrollment
5. Ongoing treatment with immune suppression for prophylaxis or treatment of GVHD including high dose steroids (e.g. prednisone > 0.25mg/kg)

TREATMENT

Inclusion Criteria:

1. Diagnosis of primary refractory or relapsed Acute Myeloid Leukemia (AML) with the exception of acute promyelocytic leukemia (APL). Patients with targetable mutations should have failed or be ineligible for targeted therapies (e.g. FLT3 inhibitors, IDH inhibitors, or anti-CD33 drug conjugate). AND patients should be suitable for consideration of allogeneic Hematopoietic Stem Cell Transplant with confirmation of an identified eligible donor by a FACT accredited transplant center and with confirmation that the center plans to proceed with transplant if CLL-1.CAR treatment induces a response they consider adequate to proceed to allogeneic HSCT.
2. CLL-1 positive tumor with at least 30% CLL-1 blasts by flow cytometry or immunohistochemistry (tissue) assessed by a CLIA certified Flow Cytometry/Pathology laboratory
3. Age ≤75 years NOTE: The first six (6) patients treated on the study will be adults (≥18 yrs of age).
4. AST/ALT less than 5 times the upper limit of normal
5. Bilirubin less than 3 times the upper limit of normal
6. Estimated GFR ≥ 60ml/min
7. Pulse oximetry of > 92% on room air
8. Karnofsky/Lansky ≥ 60
9. No systemic chemotherapy at least 2 weeks prior to treatment on study and must be recovered from all acute toxic effects of prior chemotherapy at time of treatment
10. Available autologous transduced activated peripheral blood T-cell product with ≥ 20% expression of CLL-1.CAR.28z by flow cytometry
11. Life expectancy > 12 weeks
12. Sexually active patients must be willing to utilize one of the more effective birth control methods during the study and for 6 months after the study is concluded. The male partner should use a condom
13. Informed consent explained to, understood by, and signed by patient/guardian. Patient/guardian given copy of informed consent.

Exclusion Criteria:

1. Diagnosis of acute promyelocytic leukemia (APL)
2. Currently receiving any investigational agents or having received any tumor vaccines within the previous 6 weeks.
3. History of hypersensitivity reactions to murine protein-containing products.
4. Pregnant or lactating.
5. Active infection with HIV or HTLV.
6. Clinically significant bacterial, viral or fungal infection requiring ongoing antifungal therapy without improvement,.
7. Fever of unknown origin without complete work-up including imaging (CT head, sinus, chest, abdomen/pelvis)
8. Cardiac criteria: Prolonged QTc with maximum interval as defined by age; Uncontrolled atrial fibrillation/flutter; Myocardial infarction; Cardiac echocardiography with LVSF<30% or LVEF<50% or clinically significant pericardial effusion; Cardiac dysfunction NYHA III or IV; Confirmation of absence of these conditions within 6 months of treatment.
9. CNS abnormalities: Presence of CNS disease defined as detectable cerebrospinal blast cells in a sample of CSF with ≥ 5 WBCs per mm^3 or chloroma on imaging, History or presence of an underlying CNS disorder such as a seizure disorder requiring current use of antiepileptic medications, cerebrovascular ischemia/hemorrhage within prior 6 months, dementia, cerebellar disease, or any autoimmune disease with CNS involvement.
10. Use of serotherapy with Campath or Anti-Thymocyte Globulin (ATG) within the last 28 days
11. Use of Donor Lymphocyte Infusion (DLI) or other cellular therapy product within 30 days
12. Acute GVHD ≥ Grade 2 or moderate to severe (formerly extensive) chronic GVHD
13. Administration of high dose steroids >1 mg/kg within the preceding 5 days or currently receiving > 0.25 mg/kg of Prednisone equivalent
14. Hyperleukocytosis (WBC ≥50K) or rapidly progressive disease that in the estimation of the investigator would compromise the ability of the patient to complete the study.

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2020-07-09 (Actual); Primary Completion 2025-03-24 (Actual); Study Completion 2038-07-31 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) rate | 4 weeks post T cell infusion
  To assess dose limiting toxicities per protocol-defined CLL-1.CAR T related adverse events and CTCAE v5.0

SECONDARY OUTCOMES:
Overall Response Rate | 4 weeks post T cell infusion
  To measure the anti-tumor effects of CLL-1.CAR T-cells in patients with acute myeloid malignancies.

CONTACTS AND LOCATIONS:
Overall Officials: LaQuisa Hill, MD, Principal Investigator — Cell and Gene Therapy, Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No